CLINICAL TRIAL: NCT04424745
Title: A Feasibility Study of Transcranial Direct Current Stimulation with Attention Bias Modification Training for Binge Eating Disorder
Brief Title: Neuromodulation with Attention Bias Modification Training for Binge Eating Disorder
Acronym: TANDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TANDEM01
Record Dates: First submitted 2020-05-26; First posted 2020-06-11 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-06

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attention Bias Modification Training with real tDCS (Active Comparator)
  Interventions: Other: Simultaneous Attention Bias Modification Training and Transcranial Direct Current Stimulation (tDCS)
- Attention Bias Modification Training with sham tDCS (Placebo Comparator)
  Interventions: Other: Simultaneous Attention Bias Modification Training and Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Other: Simultaneous Attention Bias Modification Training and Transcranial Direct Current Stimulation (tDCS) — Participants will receive 10 sessions of computerised attention bias modification training with either real or sham tDCS. Participants will self-administer tDCS at home, with research supervision, and complete attention bias modification training on a laptop or desktop computer while receiving stimulation. Sessions will be completed week daily for 2-3 weeks.

SUMMARY:
Binge eating disorder (BED) is a common and disabling eating disorder (ED) which has significant effects on psychological wellbeing, physical health, and quality of life. Talking therapies, most notably cognitive behaviour therapy (CBT), are presently recommended for the treatment of BED. However, outcomes from treatment are inadequate. Therefore, there is a need for development of new treatments.

This study aims to investigate the feasibility of combining Attention Bias Modification Training (ABMT) and Transcranial Direct Current Stimulation (tDCS) to reduce binge-eating behaviour and craving for food in people with BED.

ABMT is a computerised training that seeks to alter responses towards food that people are not consciously aware of. During ABMT, participants are trained to 'look towards' low-calorie food and 'look away' from high-calorie food. TDCS is a safe, well tolerated, non-invasive form of brain stimulation which is suitable for supervised self-administration. It stimulates specific brain areas using a mild electrical current (2 mA) via small electrodes placed on the scalp. In this study, participants will be randomly allocated to receive either ABMT with real tDCS or ABMT with sham tDCS. ABMT and real/sham tDCS will be delivered simultaneously, i.e. participants will engage in ABM training whilst receiving tDCS. All participants will be remotely supervised by the study researcher for the duration of each treatment session.

Biological male and female adults (aged 18-60) of any gender will be eligible to take part if they have a DSM-V of BED and they are overweight or obese.

Taking part will involve completing 10 sessions of combined ABMT and real or sham tDCS over 2-3 weeks. Binge frequency, food craving and other outcomes will be measured at the start of the study, end of the study, and at the 6-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese according to WHO criteria (BMI>25 kg/m²)
* Meet criteria for full-syndrome DSM-5 Binge Eating Disorder (BED)
* Right-handed
* Must use and understand English as a language for everyday conversation
* Access to a laptop or desktop computer with webcam

Exclusion Criteria:

* Visual impairments that cannot be corrected with contact lenses or glasses
* Pregnancy
* History of neurological disease and/or seizure
* Having any metallic implants anywhere in the head or body
* History of head or eye injury
* Significant health problems in the previous six months
* Lifetime diagnosis of substance dependence, psychosis, bipolar disorder, borderline personality disorder
* Other primary psychiatric disorder requiring treatment in its own right
* Taking psychotropic medication other than a stable dosage of selective serotonin reuptake inhibitors (SSRI) for at least 14 days prior to study enrollment
* Adults consuming more than 14 units of alcohol per week who are unwilling to reduce their alcohol intake for the duration of the treatment.
* Current illicit drug use.
* Learning difficulties that would preclude safe tDCS self-administration and/or completion of questionnaire measures and neurocognitive tasks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Achievement of a 'steady state' of recruitment | Start of Recruitment to 12 months
  Recruitment rate/month over months will be assessed to demonstrate that recruitment targets for the main trial can be met within an adequate time-frame. An average of 3 patients per month must be recruited (randomised) over a consecutive 12 month period (a minimum of 36 patients) in order to demonstrate a 'steady state' of recruitment.

SECONDARY OUTCOMES:
Eating Disorder Symptoms | Baseline to 6 week follow up (on average, 8 weeks after baseline assessment)
  The Eating Disorder Examination Questionnaire (EDE-Q) will be used to assess eating disorders symptoms. The EDE-Q is a 36-item self-report quesitonnaire, and a higher global score indicates more severe eating disorder symptoms.
Craving for food | Baseline to 6 week follow up (on average, 8 weeks after baseline assessment)
  The Food Craving Questionnaire (FCQ) will be used to assess trait-level craving for food. Total scores can range between 15 and 90, with higher scores indicating more frequent and intense food cravings.
General psychopathology | Baseline to 6 week follow up (on average, 8 weeks after baseline assessment)
  The Depression, Anxiety and Stress- Scale (DASS-21) is a 21-item self-report questionnaire which aims to evaluate mood, anxiety and stress levels over the previous week. Sum scores for the total DASS range between 0 and 120, with higher scores indicating more severe psychopathology. Sub-scales assess depression, anxiety and stress symptoms specifically, and scores range from 0 to 42, with higher scores indicating more severe symptoms.
Physical Health | Baseline to 6 week follow up (on average, 8 weeks after baseline assessment)
  Weight and height will be combined to report body mass index in kg/m^2
Food related attention | Baseline to 6 week follow up (on average, 8 weeks after baseline assessment)
  The Food Attention Network Task (Food-ANT) will be used to assess three components of attention (i.e. orienting, alerting and executive function) using food (low- and high-calorie) versus non-food pictures (neutral items). Change in reaction time will be used to assess change in orienting, alerting and executive function.
Attention Bias for Food | Baseline to 6 week follow up (on average, 8 weeks after baseline assessment)
  The Visual Probe Task (VP) will be used to assess visuo-spatial attention biases for food cues. Change in dwell time measured by eye tracking and reaction time will be used to assess change in attention bias for food cues.
Working Memory | Baseline to post treatment (on average 18 days after baseline assessment)
  Participants are presented with a continuous stream of stimuli (either faces or words), and for every stimulus, the participant must indicate (yes/no) whether or not the current stimulus is the same as the one presented three trials back. This is known as the N-Back and is a measure of working memory. Higher numbers of correct responses indicates superior working memory function.
Face Affective Go/No Go | Baseline to post treatment (on average 18 days after baseline assessment)
  Neuropsychological task measuring information processing biases for positive and negative facial expressions. The participant is told a target emotion and asked to press a button only when the target emotion is present. The task consists of six blocks, each of which presents a series of faces showing either the target emotion or a differently valenced distractor. Reaction times are calculated for correct responses for each condition. Affective bias scores are calculated by subtracting the sad target/happy distractor condition reaction time from the happy target/sad distractor condition reaction time.
Cognitive Flexibility | Baseline to post treatment (on average 18 days after baseline assessment)
  In Wisconsin Card Sorting Test (WCST) participants are asked to sort 64 cards to match either color (red, blue, yellow, or green), form (crosses, circles, triangles, or stars), or number of figures (one, two, three, four). During the task, the sorting rule changes discreetly from color to form or number of figures without the participants being informed. The participants have to shift sets accordingly and sort cards following the new sorting rule. Set shifting difficulties are indicated by preservative errors; thus, higher scores on this test represent poorer cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Schmidt, MD PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No